CLINICAL TRIAL: NCT03630211
Title: Autologous Stem Cell Transplantation With CD34-Selected Peripheral Blood Stem Cells (PBSC) in Patients With Treatment Resistant Systemic Sclerosis (SSc)
Brief Title: Autologous Stem Cell Transplantation in Patients With Systemic Sclerosis
Acronym: SSc
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Paul Szabolcs (Other)
Responsible Party: Sponsor-Investigator, Paul Szabolcs, Chief, Division of Blood and Marrow Transplantation and Cellular Therapy, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY19050297
Record Dates: First submitted 2018-08-07; First posted 2018-08-14 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Systemic Sclerosis; Diffuse Sclerosis Systemic; Interstitial Lung Disease; Pulmonary Hypertension
Keywords: Stem Cell Transplantation; Systemic Sclerosis; Scleroderma; Interstitial Lung Disease; ILD (Interstitial Lung Disease); Pulmonary Hypertension; BMT ( bone marrow transplantation); Autologous
MeSH Terms: conditions — Scleroderma, Systemic; Scleroderma, Diffuse; Lung Diseases, Interstitial; Hypertension, Pulmonary | interventions — Cyclophosphamide; Mesna; Rituximab; Alemtuzumab; Thiotepa; Granulocyte-Macrophage Colony-Stimulating Factor; Filgrastim; Immunoglobulins, Intravenous; Whole-Body Irradiation; Antilymphocyte Serum; thymoglobulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Autologous Stem Cell Transplantation (Experimental): CD34-selected autologous stem cell being performed on CliniMACS depletion device. Conditioning regimen will not start sooner than 3 weeks, and ideally no more than 90 days, after cyclophosphamide dose in the mobilization regimen.
  Interventions: Drug: Cyclophosphamide; Drug: Mesna; Drug: Rituximab; Drug: Alemtuzumab; Drug: Thiotepa; Drug: GM-CSF; Drug: Intravenous immunoglobulin; Radiation: Total Body Irradiation; Drug: Anti Thymocyte Globulin

INTERVENTIONS:
Drug: Cyclophosphamide — Stem Cell Mobilization
Drug: Mesna — Stem Cell Mobilization
Drug: Rituximab — Transplantation Conditioning
  Other Names: Rituxan
Drug: Alemtuzumab — Transplantation Conditioning
  Other Names: Campath-1H
Drug: Thiotepa — Transplantation Conditioning
Drug: GM-CSF — Transplantation Conditioning
  Other Names: Neupogen, Filgrastim
Drug: Intravenous immunoglobulin — Transplantation Conditioning
Radiation: Total Body Irradiation — Transplantation Conditioning
Drug: Anti Thymocyte Globulin — Transplantation Conditioning
  Other Names: Thymoglobulin

SUMMARY:
The purpose of this study is to determine whether a regimen of high-dose immunoablative therapy will demonstrate safety that is consistent or improved with other published regimens in SSc patients, while maintaining a treatment effect.

DETAILED DESCRIPTION:
This is a single center, phase II trial where after a process of stem cell mobilization and conditioning, subjects receive a CD34-selected autologous peripheral blood stem cell rescue. By virtue of positive selection for the stem/progenitor cell marker of CD34, the graft will be depleted for T, B and NK lymphocytes and other immune cells such as monocytes that may be pathogenic. This is an open label study and there will be no randomization or blinding as a part of this study.

The proposed regimen of high-dose immunoablative therapy will demonstrate safety that is consistent or improved with other published regimens in SSc patients, while maintaining a treatment effect.

The primary objectives of this study are to determine the safety and treatment effect of high-dose immunoablative therapy followed by transplantation of CD34+ positively selected peripheral blood stem cells (PBSC) for systemic scleroderma (SSc) patients using a regimen designed to maximize patient safety while also aiming to eradicate autoreactive clones responsible for the disease. Safety will be determined by monitoring for death of any cause, and severe or life-threatening infections. Treatment effect will be determined by assessing event-free survival in comparison to a SSc observational cohort control group treated with standard of care medication (mycophenolate mofetil) at 12 and 36 months post hematopoietic stem cell transplant (HSCT). Enrolled subjects will be followed for survival, secondary malignancies, and SSC activity at least yearly up to 36 months post-HSCT.

The secondary objectives of this study are to:

* To assess cutaneous disease response to high dose immunosuppressive therapy (HDIT) by comparing pre- and post-transplant measurements of the modified Rodnan skin score (mRSS).
* To assess pulmonary disease response by longitudinally tracking FVC (pulmonary function test) and DLCO (diffusing capacity of the lung for carbon monoxide) yearly up to 36 months post-HSCT.
* To evaluate the treatment effect on disease activity/progression, as indicated by severity measures of cardiac, pulmonary, musculoskeletal, gastrointestinal, vascular and renal organ involvement, and need for concomitant disease-modifying antirheumatic drugs (DMARD) use.
* To evaluate quality of life by comparing pre- and post-transplant quality of life measurements. These measurements will include the Scleroderma Health Assessment Questionnaire (SHAQ), the Medical Outcomes Study Questionnaire Short Form 36 Health Survey (SF-36) and the Scleroderma Skin Patient Reported Outcome (SSPRO) pre- and post-mobilization.

ELIGIBILITY:
Cohort 1: Children, Adolescents and Young Adults (Cohort 1)

Inclusion:

Individuals must meet all the following criteria to be eligible for this study.

1. Patient, parent, or legal guardian must have given written informed consent. For patients ≥ 168 years of age who are developmentally able, assent or affirmation will be obtained.
2. Age 8-24, inclusive, at time of consent.
3. Diagnosed with Systemic Sclerosis (SSc) at the age of ≤19.
4. Failure to respond, specifically no improvement or progression of disease, to at least 2 disease-modifying antirheumatic drugs (DMARDS) within 12 months of consent with any of the following conditions:

   1. Progression of skin thickening over the past 6 months or Modified Rodnan skin score (mRSS) ≥ 20
   2. Progression of ILD within 18 months prior to consent. Progression to be determined by either of the following:

      * CT scan showing increased ground glass opacities or reticulations OR
      * Pulmonary function testing (PFTs) showing a decrease in FVC% or DLCO% predicted value of ≥10%.
   3. Myositis - CPK > 2x upper limit of normal or MRI consistent with myositis
   4. Childhood Myositis Assessment Score < 30
   5. Arthritis
   6. Digital tip ulcerations
5. Cardiology clearance to undergo stem cell transplantation (documented in subject's medical chart)
6. Negative for human immunodeficiency virus (HIV), hepatitis B virus and hepatitis C virus, all confirmed by PCR testing.
7. Negative pregnancy test for females. who have reached menarche.

87. All females of childbearing potential and sexually active males must agree to use an FDA approved method of birth control for up to 24 months after BMT or for as long as they are taking any medication that may harm a pregnancy, an unborn child or may cause a birth defect.

Exclusion:

Individuals who meet any of these criteria are not eligible for this study.

1. FVC <35%, determined by pulmonary function tests for those able to complete spirometry adequately (per investigator's determination)
2. O2 sat <92% at rest in room air
3. Estimated CrCl <40 mL/min,using Cockcroft-Gault formula based on actual body weight.
4. Active, untreated SSc renal crisis at the time of consent.
5. ALT > 4x upper limit of normal.
6. Active, uncontrolled infection that would be a contraindication to safe use of high-dose immunosuppressive therapy or cyclophosphamide.
7. Hematologic abnormalities as defined by any of the following peripheral blood counts:

   1. ANC < 1500 cell/µL.
   2. Platelets < 100,000 cells/ µL.
   3. Hemoglobin < 9.0 g/dL.
8. Malignancy within 2 years prior to enrollment, excluding adequately treated squamous cell cancer, basal cell carcinoma or carcinoma in situ. Treatment should have been completed with cure/remission status documented for at least 2 years.
9. Past or current medical problems or findings from medical history, physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Cohort 2 for Adults

Inclusion:

Individuals must meet all the following criteria to be eligible for this study.

1. Patient, parent, or legal guardian must have given written informed consent. For patients ≥ 16 years of age who are developmentally able, assent or affirmation will be obtained.
2. Age 1618-705560, inclusive, at time of consent. Patients up to age 24, diagnosed with SSc at age ≤ 19, will be included in Cohort 1 and evaluated according to the Pediatric and Young Adult criteria listed in sections 3.1.1 and 3.1.2.
3. Diagnosed with Systemic Sclerosis (SSc), according to the 2013 ACR/EULAR criteria (van den Hoogen et al., 2013).
4. All patients must meet either the following skin or ILD criteria. Disease duration is defined as time from first non-Raynaud symptom.

   Skin Criteria: Diffuse SSc, defined by presence of proximal skin thickening and:

   A. If disease duration is of <2 years, patients must have a calculated mortality risk prediction score which places them in the intermediate or high- risk category (Domsic et al., 2016). Refer to Appendix 5 for calculation criteria.

   B. If disease duration is of >2 years, patients must have evidence of active cutaneous disease based upon 1) a worsening Modified Rodnan Skin Score (MRSS) in the preceding three months or 2) the presence of palpable tendon friction rubs.

   ILD Criteria:

   A. The presence of recognized fibrosis on imaging of <2 years AND either > 10% of lung involvement by CT scan or FVC% pred <80% or B. Fibrosis on imaging of any duration with a decline in FVC% pred of ≥10% over the preceding 12-18 months.
5. Negative for human immunodeficiency virus (HIV), hepatitis B virus and hepatitis C virus, all confirmed by PCR testing.
6. Negative pregnancy test for females.
7. All females of childbearing potential and sexually active males must agree to use an FDA approved method of birth control for up to 24 months after BMT or for as long as they are taking any medication that may harm a pregnancy, an unborn child or may cause a birth defect.

Exclusion Criteria Individuals who meet any of these criteria are not eligible for this study.

1. Moderate to severe cardiac involvement defined by any of the following:

   1. New York Heart Association classification of heart failure ≥3.
   2. Left ventricular ejection fraction (LVEF) <50% as determined by cardiac MRI.
   3. Significant pulmonary hypertension, for subjects ≥ 18 years of age, defined as mean PASP ≥30 mmHg determined by right heart catheterization, or for subjects ≤ 17 years of age, defined as mean PASP >45 mmHg, determined by echocardiogram.
   4. Atrial tachycardia, atrial fibrillation or atrial flutter of ≥1-minute duration, determined by electrocardiogram (EKG) or, cardiac event monitor and/or implanted loop recorder (if applicable), or on anti-arrhythmic therapy for the arrhythmias listed above.
   5. Ventricular tachycardia of ≥6 beats at rate of ≥100 beats per minute, determined by EKG or, cardiac event monitor and/or implanted loop recorder (if applicable), or on an anti-arrhythmic therapy for any ventricular arrhythmia.
   6. Left bundle branch block, bifascicular heart block, Mobitz 2 heart block, complete heart block or infarction pattern as determined by EKG or, cardiac event monitor and/or implanted loop recorder
   7. Presence of pacemaker or implantable cardioverter defibrillator.
2. Moderate to severe pulmonary involvement defined by any of the following:

   1. Hemoglobin-corrected DLCO <45%, determined by pulmonary function tests.
   2. FVC <45%, determined by pulmonary function tests.
   3. pO2 <70 mmHg, determined by an arterial blood gas (not applicable for subjects ≤17 years of age).
   4. pCO2 ≥45 without supplemental O2 determined by an arterial blood gas (not applicable for subjects ≤17 years of age).
   5. O2 sat <92% at rest without supplemental O2, determined by an arterial blood gas (not applicable for subjects ≤17 years of age).
   6. Six-minute walk (6MW) results <400 feet.
3. Steroid therapy defined by either of the following:

   1. Subjects who received > 10 mg/day prednisone or equivalent within 30 days prior to start of conditioning regimen on Day -21.
   2. Subjects who have been treated for concurrent illnesses (eg, asthma) with the equivalent of prednisone 1 mg/kg/day or its equivalent for > 5 days on > 2 occasions during the previous 12 months (prior to conditioning) or > 1 occasion in the prior 6 months (prior to conditioning).
4. Estimated CrCl <40 mL/min,using Cockcroft-Gault formula based on actual body weight.
5. Serum creatinine >2.0 mg/dL.
6. Active, untreated SSc renal crisis at the time of consent.
7. Dependence on nutritional supplementation/hyperalimentation.
8. Active gastric antral vascular ectasia (GAVE), defined by a decrease in hemoglobin greater than 1 g/dL in the preceding 60 days, attributed to GAVE.
9. Active hepatitis defined by any of the following:

   1. AST > 2x upper limit of normal.
   2. ALT > 2x upper limit of normal.
   3. Bilirubin >2x upper limit of normal.
10. Evidence of moderate to severe periportal fibrosis, determined by liver biopsy, if applicable.
11. Active, uncontrolled infection that would be a contraindication to safe use of high-dose immunosuppressive therapy or cyclophosphamide.
12. Hematologic abnormalities as defined by any of the following peripheral blood counts:

    1. ANC < 1500 cell/µL.
    2. Platelets < 100,000 cells/ µL.
    3. Hemoglobin < 9.0 g/dL.
13. Evidence of myelodysplasia (MDS), confirmed by bone marrow aspirate, if applicable.
14. Malignancy within 2 years prior to enrollment, excluding adequately treated squamous cell cancer, basal cell carcinoma or carcinoma in situ. Treatment should have been completed with cure/remission status documented for at least 2 years, with the exception of hormonal therapy for breast cancer.
15. Females who are pregnant or who are lactating.
16. Tobacco use, by subject admission, within previous 4 weeks of time of consent.
17. History of sensitivity to murine proteins or E. coli proteins.
18. Known history of substance abuse, determined by medical record or subject admission, within 6 months of time of consent.
19. Patient with systemic reaction to anti-thymocyte globulin or any other equine gamma globulin preparation
20. Past or current medical problems or findings from physical examination or laboratory testing that are not listed above, which, in the opinion of the investigator, may pose additional risks from participation in the study, may interfere with the participant's ability to comply with study requirements or that may impact the quality or interpretation of the data obtained from the study.

Ages: 8 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Estimated)
Dates: Start 2018-07-31 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
High Dose Immunoablative therapy-Safety | Up to 36 months post HSCT
  Safety will be determined by monitoring for death of any cause, regimen-related toxicities, and severe or life-threatening infections.
Death | Post Transplant through study completion, an average of 36 months
  How many, if any, patients die
Respiratory Failure | Post Transplant through study completion, an average of 36 months
  defined by one of the following 3 criteria without explanation for causation other than disease progression: 1. decline in DLCO of ≥30% or FVC≥20% as measured by actual difference in percent predicted units; 2. Resting arterial p02 < 60 mmHg or pCO2 > 50 mmHg supplemental oxygen;3. Resting pulse oximetry of 88% or lower measured by forehead probe.
Renal Failure | Post Transplant through study completion, an average of 36 months
  Defined by chronic dialysis for >6 months or renal transplantation
The occurrence of cardiomyopathy | Post Transplant through study completion, an average of 36 months
  confirmed by clinical congestive heart failure (New York Heart Association) or LVEF (left ventricular ejection fraction) <30% on echocardiogram
Treatment-related mortality (TRM) | Mobilization through study completion, an average of 36 months
  defined as death occurring at any time after stem cell mobilization and definitely or probably resulting from treatment given in the study. TRM will be determined yearly with a focus on the first 2 years.
High Dose Immunoablative therapy-Treatment Effect | up to 36 months post HSCT (hematopoietic stem cell transplantation)
  Treatment effect will be determined by assessing event-free survival in comparison to a SSc observational cohort control group treated with standard of care medication (mycophenolate mofetil) at 12 and 36 months post hematopoietic stem cell transplant (HSCT).

SECONDARY OUTCOMES:
An increase of mRSS (modified Rodnan skin score ) by ≥5 points for skin score | Disease response will be defined as subject improvement. This will be assessed for both skin and interstitial lung disease at 12 and 24 months post-HSCT.
  To assess cutaneous response the modified Rodnan skin score (mRSS) will be used.
Increase by ≥25% if the baseline mRSS > 20. | Disease response will be defined as subject improvement. This will be assessed for both skin and interstitial lung disease at 12 and 24 months post-HSCT.
  To assess cutaneous response the modified Rodnan skin score (mRSS) will be used.
Worsening of > 10% of FVC (pulmonary function testing) | 1 year post transplant through study completion, an average of 36 months
  to evaluate interstitial lung disease an increase of ≥15% in DLCO or ≥10% of FVC (actual change in % predicted units from baseline) sustained for ≥3 months on 2 determinations.
Decrease in DLCO sustained for 3 months or longer on pulmonary function tests (PFT) | 1 year post transplant through study completion, an average of 36 months
  to evaluate interstitial lung disease an increase of ≥15% in DLCO or ≥10% of FVC (actual change in % predicted units from baseline) sustained for ≥3 months on 2 determinations.
Worsening of cardiac involvement | Post Transplant through study completion, an average of 36 months
  With use of Imaging, EKG, Echocardiogram, Cardiac MRI, right heart cauterization, implanted loop recorder and 2 week cardiac event monitor. Defined as new or worsening arrhythmias that require medical treatment of 3 months or longer, or require ablative therapy, pacemaker or defibrillator insertion or defined as a decline in ejection fraction of ≥10 EF units, determined by echocardiogram.
Development of scleroderma renal crisis (hypertensive or non-hypertensive) | Post Transplant through study completion, an average of 36 months
  Hypertensive renal crisis can be defined as a rise in SBP ≥ 30 points or DBP ≥ 20 points from baseline and one of the following: 1) Increase in baseline serum creatinine of ≥ 50%, 2) thrombocytopenia < 100,000 plts/mm3 or 3. hemolysis by blood smear or increased reticulocyte count.

CONTACTS AND LOCATIONS:
Overall Officials: Paul Szabolcs, MD, Principal Investigator — University of Pittsburgh
Locations (2):
- United States (2):
  - Children's Hospital of Pittsburgh of UPMC, Pittsburgh, Pennsylvania
  - University of Pittsburgh Medical Center, Pittsburgh, Pennsylvania

IPD SHARING:
Plan to Share IPD: No